CLINICAL TRIAL: NCT07037602
Title: The Effect of Sexual Health Education Given to Women on Sexual Myths and Self-Consciousness: A Randomized Controlled Trial
Brief Title: Sexual Health Education Given to Women
Acronym: Sexual Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator, Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sexual Health Education
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Nursing
MeSH Terms: interventions — Sex Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): All women will be given the Personal Information Form, Sexual Myths Scale and Sexual Self-Consciousness Scale as a pre-test. No intervention will be made to the control group. After 8 weeks, the women will be reunited and given the Sexual Myths Scale and Sexual Self-Consciousness Scale as a post-test.
  Interventions: Other: No Interventions
- sexual health education (Experimental): After the Personal Information Form, Sexual Myths Scale and Sexual Self-Awareness Scale are applied as a pre-test to all women, sexual health training will be given to the women in the experimental group. The training will be given in 4 sessions over 2 weeks. Demonstration, powerpoint, feedback and brainstorming methods will be used in the training.
  Interventions: Other: Sexual Health Education

INTERVENTIONS:
Other: Sexual Health Education — After the Personal Information Form, Sexual Myths Scale and Sexual Self-Awareness Scale are applied as a pre-test to all women, sexual health training will be given to the women in the experimental group. The training will be given in 4 sessions over 2 weeks. Demonstration, powerpoint, feedback and brainstorming methods will be used in the training.
  Arms: sexual health education
Other: No Interventions — No intervention will be made.
  Arms: Control group

SUMMARY:
No study was found in the literature examining the effects of sexual health education on sexual myths and self-consciousness. The aim of the study was to investigate the effects of sexual health education on sexual myths and self-consciousness in women.

DETAILED DESCRIPTION:
Sexual myths can be defined as false, stereotyped judgments that individuals believe to be true about sexuality, are generally exaggerated, have no scientific basis, and limit the freedom to live sexuality. Sexual myths are widely seen in society and can vary between cultures and societies, and even between individuals. Especially in closed-structure societies, these myths are increasingly widespread by being passed down from generation to generation. Sexual myths can cause people to have unrealistic expectations, feel inadequate due to these expectations, and feel anxious. As a result of all these, sexual dysfunctions can occur, and the treatment process can be negatively affected in people with sexual dysfunction. If sexual self-consciousness, that is, sexuality, has not yet been discovered as a personal area, if the person's idea of what to expect from sexual contact is shaped by myths, their sexual health may deteriorate. It is known that the most important factors that pave the way for sexual myths are lack of sexual education and information, the inability to openly discuss and discuss issues related to sexuality within the family, schools or society, and the inability to benefit from sufficient scientific research and publications.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-45,
* Those who have not received sexual health education before,
* Those who speak Turkish,
* Women who volunteer to participate in the research.

Exclusion Criteria:

* Those who have been medically diagnosed with sexual dysfunction,
* Women diagnosed with a psychiatric illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Sexual Self-Consciousness Scale | 2 months
  The sexual self-consciousness scale was developed by Van Lankveld, Geijen and Sykora in 2007 and adapted to Turkish by Çelik and Çakmak in 2012. The scale determines both the sexual self-consciousness and sexual self-focus and sexual shyness levels of individuals and is presented as a measurement tool based on the principle of the individual providing information about himself/herself (self-report). The sexual self-consciousness scale, which is a 5-point Likert-type (0 Totally Disagree - 4 Totally Agree), has two sub-dimensions: sexual shyness and sexual self-focus. In these sub-dimensions, the sexual shyness sub-dimension consists of items 1-6, and the sexual self-focus sub-dimension consists of items 7-12. The scale provides both a total score for sexual self-consciousness and a score for both sub-dimensions (sexual self-focus and sexual shyness). There are no reverse-coded items in the scale. The possible score range varies between 0 and 42.

SECONDARY OUTCOMES:
Sexual Myths Scale | 2 months
  The Sexual Myths Scale (CMÖ) is a scale developed by Gölbaşı, Evcili, Eroğlu, and Bircan to determine whether individuals have sexual myths. The total Cronbach's alpha coefficient is 0.91. The scale consisting of 28 items is a Likert-type measurement tool. The scale was prepared in a way that one of the answers in the range of "1=Strongly Disagree" to "5=Strongly Agree" is marked. The sexual myths scale consists of eight dimensions. These dimensions and the questions belonging to these dimensions are; gender (1,2,3,4,5,6), sexual orientation (7,8,9,10,11), age and sexuality (12,13,14,15), sexual behavior (16,17,18), masturbation (19,20), sexual violence (21,22,23,24), sexual intercourse (25,26) and sexual satisfaction (27,28).

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided